CLINICAL TRIAL: NCT01481402
Title: Liothyronine and Heart Failure. The Long Term Effect of Liothyronine on Heart Function, Body Composition and Metabolic Status
Brief Title: Liothyronine and Heart Failure. The Long Term Effect of Liothyronine on Left Ventricular Ejection Fraction (LVEF)
Acronym: LIHFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Faber (Other)
Responsible Party: Sponsor-Investigator, Jens Faber, professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HerlevH
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2014-02

CONDITIONS: Heart Failure; Low T3 Syndrome
Keywords: Heart failure; Liothyronine; Low T3 syndrome
MeSH Terms: conditions — Heart Failure; Euthyroid Sick Syndromes | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo-liothyronine (Placebo Comparator): 3 months of placebo followed by 3 months of Liothyronine treatment.
  Interventions: Drug: Liothyronine
- Liothyronine-Placebo (Other): 3 months of Liothyronine treatment followed by 3 months of Placebo treatment.
  Interventions: Drug: Liothyronine

INTERVENTIONS:
Drug: Liothyronine — Liothyronine 40 microgram per day
  Other Names: T3
  Arms: Placebo-liothyronine
Drug: Liothyronine — 3 months of placebo followed by 3 months of Liothyronine 40 microgram per day (oral)
  Other Names: T3
  Arms: Liothyronine-Placebo

SUMMARY:
Purpose: The purpose of the study is to examine if treatment with liothyronine increases left ventricular ejection fraction (LVEF) in patients with stable, chronic heart failure.

DETAILED DESCRIPTION:
The patients are examined 3 times. At baseline, after 3 months and after 6 months.After the examination is performed, they begin the study medication while admitted at Dept. of Cardiology, Herlev Hospital, for cardiac monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable, chronic systolic heart failure
* T3 ≤1.4 nmol/l in two blood samples, TSH is to be normal
* LVEF ≤ 45 % on prior echocardiography

Exclusion Criteria:

* Established thyroid illness
* Atrial fibrillation/flutter
* More than 20% ventricular extrasystoles
* Severe chronic obstructive lung disorder
* Pregnancy. Pregnancy testing will be done for fertile women
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
left ventricle ejection fraction | 3 months
  The effect of liothyronine treatment in low dose in 3 months on LVEF.

SECONDARY OUTCOMES:
Body composition | 3 months
  The effect of 3 months low dose liothyronine treatment on body composition in patients with heart failure.
Quality of Life, questionaire | 3 months
  The effect of 3 months low dose liothyronine treatment on quality of life, assessed by SF-36 and Minnesota Living with Heart Failure questionnaires in patients with heart failure.
YKL-40, YNF-alpha, hsCRP and IL-6 | 3 months
  The effect of 3 months low dose liothyronine treatment on low grade inflammation assessed by measurement of pro-inflammatory markers in patients with heart failure.
RBP 4, HBA1C, adiponectin (high and low weight), glucose and HOMA-1 | 3 months
  The effect of 3 months low dose liothyronine treatment on metabolic status in patients with heart failure.
GDF 8, SHBG, CK and PINP | 3 months
  The effect of 3 months low dose liothyronine treatment on the extrathyroidal thyroid effect in patients with heart failure.
NT-proBNP, EDV and ESV | 3 months
  The effect of 3 months low dose liothyronine treatment on heart function in patients with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Faber, MDSci, Study Director — Herlev Hospital, Dept. of Endocrinology
Locations (1):
- Herlev Hospital, Dept. of Endocrinology, Herlev, Denmark